CLINICAL TRIAL: NCT02225223
Title: Evaluation of Targeted Radiofrequency Ablation and Vertebral Augmentation Prior to or Following Radiation Therapy to Treat Painful Metastatic Vertebral Body Tumor(s) [The STARRT Study]
Brief Title: Evaluation of t-RFA and RF-TVA Prior to/Following Radiation Therapy to Treat Painful Metastatic Vertebral Body Tumor(s)
Acronym: STARRT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty Enrolling
Sponsor: Merit Medical Systems, Inc. (Industry)
Collaborators: DFINE Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DF-14-01
Record Dates: First submitted 2014-08-21; First posted 2014-08-26 (Estimated); Results first posted 2021-07-21 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-07

CONDITIONS: Metastatic Lesions in Vertebral Bodies
Keywords: metastatic lesions; vertebral body; ablation; radiation; targeted radio-frequency ablation; radio-frequency targeted vertebral augmentation; radiofrequency kyphoplasty; spine; vertebral augmentation; kyphoplasty; spinal ablation; pain; quality of life; spinal tumors
MeSH Terms: conditions — Pain; Spinal Cord Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No previous Radiation Therapy (Other): Targeted radio-frequency ablation using the STAR™ Tumor Ablation System and vertebral augmentation using the StabiliT® Vertebral Augmentation System.
  Interventions: Device: STAR™ Tumor Ablation System; Device: StabiliT® Vertebral Augmentation System
- Failed/Refuse further Radiation Therapy (Other): Targeted radio-frequency ablation using the STAR™ Tumor Ablation System and vertebral augmentation using the StabiliT® Vertebral Augmentation System.
  Interventions: Device: STAR™ Tumor Ablation System; Device: StabiliT® Vertebral Augmentation System

INTERVENTIONS:
Device: STAR™ Tumor Ablation System — Targeted-radiofrequency ablation (t-RFA)
Device: StabiliT® Vertebral Augmentation System — Radiofrequency-targeted vertebral augmentation (RF-TVA)

SUMMARY:
The purpose of this study is to evaluate treating painful metastatic lesions in vertebral bodies with pathologic fractures with targeted radiofrequency ablation (t-RFA) and vertebral augmentation (VA) prior to or following radiation therapy.

DETAILED DESCRIPTION:
Prospective, multi-center clinical study. Stratification scheme: 'Failed/Refused Further RT' and "No Previous RT"

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patient is ≥ 18 years old,
2. One to two painful vertebrae (T1-L5) with evidence of osteolytic or mixed lytic and blastic metastatic lesion by cross sectional imaging and pathologic fracture (presence of non-painful vertebrae with metastatic lesions in addition to the painful index vertebrae are allowed)
3. Never received radiation therapy at index level(s) (following consult with radiation oncologist re: conventional treatment options) OR Received radiation therapy without adequate relief from metastatic bone pain as determined by the patient and treating physician, their treating physician would not prescribe additional radiation treatments, or refuse additional radiation therapy,
4. Brief Pain Inventory (BPI) worst pain score of ≥ 4 (irrespective of medication),
5. Woman of potential childbearing age agrees to a medically effective birth control method,
6. Life expectancy of ≥ 2 months,
7. Sufficient mental capacity to comply with the protocol requirements,
8. Understands the potential risks and benefits of study participation and is willing to provide written informed consent.

Exclusion Criteria:

1. Primary tumors of the bone (e.g., osteosarcoma) at site of index vertebra(e),
2. Benign tumors of the bone (e.g. osteoid osteoma) at site of index vertebra (e),
3. Lesions due to hematologic malignancy (e.g. multiple myeloma at site of the index vertebra (e),
4. Compromise in the posterior column of the vertebral body or walls of pedicles.
5. Extra-osseous extension of metastatic lesion is >10mm,
6. Nonreversible or uncorrectable coagulopathy. INR should not be >1.5,
7. Platelet count of < 50,000 ,
8. Radiation therapy was completed on the index vertebra(e) ≤ 28 days before enrollment,
9. Change in chemotherapy agent is planned 7 days before or after enrollment (change in dose(s) permitted),
10. Index vertebra(e) had previous spine surgery including vertebroplasty or kyphoplasty,
11. Additional non-kyphoplasty/vertebroplasty surgical treatment is required for the index vertebra(e),
12. Spinal cord compression or canal compromise requiring decompression,
13. Major surgery of the spine in same region as the index vertebra(e) was performed within 3 months before enrollment,
14. Major elective surgery to the spine in same region as the index vertebra(e) is planned within 1 month following the ablation and cement procedure,
15. Requires upper and lower limb surgery that will affect functional outcomes,
16. Significant clinical morbidities (aside from the index vertebra(e) and recurrent cancer) that may interfere with data collection that affects pain and functional results,
17. Medical/surgical conditions contrary to the kyphoplasty procedure (e.g., presence of active or incompletely treated local infection, severe pulmonary insufficiency),
18. Bedridden due to paralysis or neurological decline,
19. Currently pregnant or nursing, or planning pregnancy (in the period up to 6 months) following the index procedure(s),
20. Known allergy to bone cement,
21. Has a heart pacemaker or other electronic device implants
22. Concurrent participation or participation within the last 30 days prior to enrollment in any clinical trial with an investigational medicinal drug/chemotherapeutic or biologic or medical product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-12; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack Jennings, MD, Principal Investigator — Washington University School of Medicine
Locations (14):
- United States (14):
  - USC, Los Angeles, California
  - Torrance Memorial Medical Center, Torrance, California
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Feinberg School of Medicine, Chicago, Illinois
  - Vascular and Interventional Radiology, La Grange, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mayo Clinic, Rochester, Minnesota
  - Washington University/Siteman Cancer Center, St Louis, Missouri
  - Wake Forest, Winston-Salem, North Carolina
  - University of Texas Southwestern, Dallas, Texas
  - St. Marks Hospital, Salt Lake City, Utah
  - Inova Alexandria Hospital, Alexandria, Virginia
  - Providence Sacred Heart, Spokane, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | No Previous Radiation Therapy | Failed/Refuse Further Radiation Therapy
Started | 27 | 8
Completed | 8 | 3
Not Completed | 19 | 5
Not completed — Death | 10 | 1
Not completed — Lost to Follow-up | 5 | 0
Not completed — Other | 1 | 2
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Previous Radiation Therapy | Failed/Refuse Further Radiation Therapy | Total
Number analyzed (Participants) | 27 | 8 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.1 (15.3) | 53.4 (15.23) | 60.2 (15.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 4 | 19
  Male | 12 | 4 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 26 | 8 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 4 | 6
  White | 23 | 4 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Primary Cancer [Count of Participants; unit: Participants]
  Breast Cancer | 6 | 2 | 8
  Prostate Cancer | 1 | 2 | 3
  Prostate Cancer and Other | 2 | 0 | 2
  Small Cell Lung Cancer | 2 | 0 | 2
  Non-Small Cell Lung Cancer | 2 | 1 | 3
  Thyroid Cancer | 1 | 0 | 1
  Other | 13 | 3 | 16
Brief Pain Inventory (BPI -Short Form) - 24 hour worst pain [Mean (Standard Deviation); unit: units on a scale] — The BPI asks subjects to rate pain by circling the one number that best describes pain at its worst in the last 24hrs. 0=no pain and 10=pain as bad as (you) can imagine. Results are presented in response to Q3 of the BPI only (i.e. pain at its worst in the last 24hrs). This was accomplished using the BPI short form.
  units on a scale | 7.9 (1.93) | 7.1 (1.46) | 7.7 (1.84)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Brief Pain Inventory Q3 Worst Pain Score at 6 Weeks
Description: The Brief Pain Inventory (BPI) short form rates pain on a scale from 0 to 10 (with 0=no pain and 10=worst pain you can imagine). The response is from Q3 reporting worst pain within the last 24 hours. Primary outcome is measuring the mean change from baseline in BPI worst pain score at 6 weeks.
Time Frame: Mean change from baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Previous Radiation Therapy | Failed/Refuse Further Radiation Therapy
Number analyzed (Participants) | 27 | 8
score on a scale | 2.3 (1.48) | 1.8 (1.13)

2. Secondary Outcome: Mean Change From Baseline in Brief Pain Inventory Worst Pain Score at Visits Prior to 6 Weeks
Description: Measured by Brief Pain Inventory (BPI) Pain Q3, The Brief Pain Inventory (BPI) short form rates pain on a scale from 0 to 10 (with 0=no pain and 10=worst pain you can imagine). The response is from Q3 reporting worst pain within the last 24 hours. Secondary outcome is measuring the mean change from baseline in BPI worst pain score prior to 6 weeks.
Time Frame: Mean Change from Baseline prior to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Previous Radiation Therapy | Failed/Refuse Further Radiation Therapy
Number analyzed (Participants) | 27 | 8
score on a scale | 2.1 (1.75) | 1.5 (1.24)

3. Secondary Outcome: Brief Pain Inventory Q3 Worst Pain Score by Visit
Description: The Brief Pain Inventory (BPI) short form rates pain on a scale from 0 to 10 (with 0=no pain and 10=worst pain you can imagine). The response is from Q3 reporting worst pain within the last 24 hours. Secondary outcome is the response to Q3 at Weeks 1, 2 and 6.
Time Frame: Week 1, Week 2, Week 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | No Previous Radiation Therapy | Failed/Refuse Further Radiation Therapy
Number analyzed (Participants) | 27 | 8
score on a scale
  Week 1 | 4.5 (3.00) | 4.9 (2.67)
  Week 2 | 3.9 (3.05) | 5.3 (2.12)
  Week 6 | 3.6 (2.87) | 3.8 (1.91)

ADVERSE EVENTS:
Time Frame: Adverse events were collected through time of (early) study termination due to lack of enrollment, through 6 months.
Description: All cause mortality was collected. Of 35 enrolled subjects, 9 died due to disease progression and 2 died due to other reasons (one was listed as hospice and the other as "unknown"). There were 0 participants considered to have experienced Serious Adverse Events (SAEs) and the participants who died due to disease progression and other reasons are not considered SAEs.
Arm/Group | No Previous Radiation Therapy | Failed/Refuse Further Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 10/27 | 1/8
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/8
Other Adverse Events (participants affected / at risk) | 0/27 | 0/8

LIMITATIONS AND CAVEATS:
Study was terminated due to difficulty with enrollment. Analysis of data is limited due to early termination of study and incomplete enrollment and completion of study subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No